CLINICAL TRIAL: NCT02714582
Title: Patient Participation at the Bedside: Feasibility, Appropriateness, Meaningfulness and Effectiveness of Bedside Shift Reporting. A Matched Controlled Trial
Brief Title: Feasibility, Appropriateness, Meaningfulness and Effectiveness of Bedside Shift Reporting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HA/RP/2015/086/EC; B670201627044 (Other: Ethics Committee UZ Gent)
Record Dates: First submitted 2016-02-29; First posted 2016-03-21 (Estimated); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Nursing; Bedside Shift Report; Patient Participation
Keywords: Shift report; Bedside; Nursing; Matched controlled trial; Mixed method; Patient participation
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bedside shift report (Experimental): The experimental group (nurses and patients) will:
  * develop a tailored BSR-intervention by use of co-design, diagnostic interviews, and pilot testing
  * use the tailored BSR-intervention, with participation of the patient, instead of the regular nurse shift report
  Interventions: Behavioral: Bedside shift report
- No bedside shift report (No Intervention): The control group will not use bedside shift report, but will use the regular nurse shift report without participation of the patient

INTERVENTIONS:
Behavioral: Bedside shift report — Bedside shift report is a process where shift-to-shift report between nurses is, if approved by the patient, executed at the patient's bedside in order to improve the patient's involvement (Anderson & Mangino 2006).
  Other Names: Bedside shift handover
  Arms: Bedside shift report

SUMMARY:
Hospitals face the challenge to continually improve their quality of care. In order to achieve this goal, they have to focus on both improving clinical practice and increasing the involvement of patients in the healthcare process. Both factors are equally important to quality of care. The World Health Organization highlights the role that patients and their family could play in the improvement of healthcare. Active patient participation reduces communication errors, increases patient empowerment and is associated with positive health and psychosocial outcomes. A possible strategy to improve patient participation through communication can be bedside shift report (BSR).

Bedside shift report is a process where shift-to-shift report between nurses is, if approved by the patient, executed at the patient's bedside in order to improve the patient's involvement. Bedside shift report has the potential to result in more patient satisfaction, better clinical outcomes, improvement of health education and enhanced team coherence. Preliminary research indicates that BSR decreases safety incidents and adverse events and readmissions, positively influences staff satisfaction, offers beneficial financial effects by reducing nurses' overtime, and allows direct patient care to start earlier.

Despite of these effects, rigorous and large-scale scientific research on this topic is lacking. Currently, the available evidence is scarce and mostly consists of single case or small-scale studies. Longitudinal results on effectiveness and sustainability of BSR are also unknown or inconclusive. There is a need for an increased number of controlled studies to evaluate the impact of BSR on patient, staff and economic outcomes and its longitudinal results.

The aim of this study is four-folded:

1. The development and fine-tuning of a BSR-intervention and implementation protocol by using diagnostic interviews, co-design, and pilot studies.
2. A quantitative evaluation of BSR in comparison with care as usual on patient-related, clinical, and nurse-related outcomes.
3. A qualitative evaluation of the feasibility, appropriateness and meaningfulness of BSR as a method to improve communication and patient participation with a particular interest in the experience of benefits and disadvantages by healthcare professionals and patients.
4. A process evaluation of BSR to determine the intervention fidelity and to assess the evolution of BSR over the period of the study (e.g. adaptations, consistent practice).

The study design was based on the Medical Research Council-framework for developing and evaluating complex interventions. Power calculation indicates a minimum of 5 experimental wards with 35 patients should be included in the study. The hospital, the specialization of the ward and the nurse-patient ratio will be used for the matched controlled assignment.

ELIGIBILITY:
Patients

Inclusion Criteria:

* Admitted on a participating hospital ward
* Be conscious
* Speak Dutch
* Participated in at least 3 bedside shift reports

Exclusion Criteria

* Dementia or other severe cognitive/mental disorders

Nurses

Inclusion Criteria:

* Work on a participating hospital ward
* Have at least six months of experience on the ward
* Have participated in 10 bedside shift reports or more

Exclusion Criteria:

* No hands-on patient contact
* Internship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2016-03; Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in Patient Empowerment | 24 months: 4 data collections during the study (baseline, 12 months, 18 months, 24 months)
  The change in Patient Empowerment during the study will be investigated by use of repeated measures. The patterns of change between baseline, 12 months, 18 months, and 24 months will be evaluated.
  The data will be collected by use of a questionnaire for patients. A validated tool, the Patient Activation Measure (PAM13), will be used.

SECONDARY OUTCOMES:
Change in Quality of Care | 24 months: 4 data collections during the study (baseline, 12 months, 18 months, 24 months)
  The change in Quality of Care during the study will be investigated by use of repeated measures. The patterns of change between baseline, 12 months, 18 months, and 24 months will be evaluated.
  The data will be collected by use of a questionnaire for patients. A validated tool, the QPP (Quality of care from the Patient's Perspective), will be used.
Change in Individualized Care (patient) | 24 months: 4 data collections during the study (baseline, 12 months, 18 months, 24 months)
  The change in Individualized Care during the study will be investigated by use of repeated measures. For patients, the patterns of change between baseline, 12 months, 18 months, and 24 months will be evaluated.
  The data will be collected by use of a questionnaire for patients. A validated tool, the ICS (Individualized Care Scale), will be used.
Change in Individualized Care (nurse) | 24 months: 2 data collections during the study (baseline, 24 months)
  The change in Individualized Care during the study will be investigated by use of repeated measures. For nurses, the patterns of change between baseline and 24 months will be evaluated.
  The data will be collected by use of a questionnaire for nurses. A validated tool, the ICS (Individualized Care Scale), will be used.
Change in Job Satisfaction | 24 months: 2 data collections during the study (baseline, 24 months)
  The change in Job Satisfaction during the study will be investigated by use of repeated measures. The patterns of change between baseline and 24 months will be evaluated.
  The data will be collected by use of a questionnaire for nurses. A validated tool, the MOAQ-JSS (Michigan Organizational Assessment Questionnaire - Job Satisfaction Subscale), will be used.
Change in Turnover Intention (1) | 24 months: 2 data collections during the study (baseline, 24 months)
  The change in Turnover Intention during the study will be investigated by use of repeated measures. The patterns of change between baseline and 24 months will be evaluated.
  The data will be collected by use of a questionnaire for nurses. A validated tool, the MOAQ-TIS (Michigan Organizational Assessment Questionnaire - Turnover Intention Subscale), will be used.
Change in Turnover Intention (2) | 24 months: 2 data collections during the study (baseline, 24 months)
  The change in Turnover Intention during the study will be investigated by use of repeated measures. The patterns of change between baseline and 24 months will be evaluated.
  The data will be collected by use of a questionnaire for nurses. Two questions from the RN4CAST (Nurse Forecasting: Human Resources Planning in Nursing) are used.
Change in Coordination of the Care Process | 24 months: 2 data collections during the study (baseline, 24 months)
  The change in Coordination of the Care Process during the study will be investigated by use of repeated measures. The patterns of change between baseline and 24 months will be evaluated.
  The data will be collected by use of a questionnaire for nurses. A validated tool, the CPSET-COR (Care Process Self Evaluation Tool - Coordination subscale), will be used.
Change in Communication | 24 months: 2 data collections during the study (baseline, 24 months)
  The change in Communication during the study will be investigated by use of repeated measures. The patterns of change between baseline and 24 months will be evaluated.
  The data will be collected by use of a questionnaire for nurses. A validated tool, the CPSET-COM (Care Process Self Evaluation Tool - Communication subscale), will be used.
Change in Work Interruptions (1) | 24 months: 2 data collections during the study (baseline, 24 months)
  The change in Work Interruptions during the study will be investigated by use of repeated measures. The patterns of change between baseline and 24 months will be evaluated.
  The data will be collected by use of a questionnaire for nurses. A non-validated tool to measure nurses' perceptions on work interruptions, developed by the researchers, will be used.
Change in Work Interruptions (2) | 24 months: 2 data collections during the study (baseline, 24 months)
  The change in Work Interruptions during the study will be investigated by use of repeated measures. The patterns of change between baseline and 24 months will be evaluated..
  The data will be collected from electronic databases from within the participating hospitals that measure the number of work interruptions ('calls for assistance').
Change in Patient Participation | 24 months: 2 data collections during the study (baseline, 24 months)
  The change in Patient Participation during the study will be investigated by use of repeated measures. The patterns of change between baseline and 24 months will be evaluated.
  The data will be collected by use of a questionnaire for nurses. Five questions from a validated tool, the PaCT-HCW (Patient Participation Culture Tool for Healthcare Workers), will be used.
Change in Hospital Acquired Pressure Ulcers (HAPU) | 24 months: 4 data collections during the study (baseline, 12 months, 18 months, 24 months)
  The change in incidence of HAPU's during the study will be investigated by use of repeated measures. The patterns of change between baseline, 12 months, 18 months, and 24 months will be evaluated.
  The data will be collected from the patient's medical file. The timeframe for registration is from the admission on the ward until discharge from the ward. Any HAPU's during the patient's stay on the ward on heel and sacrum will registered by use of the NPUAP/EPUAP classification system.
Change in Patient Falls | 24 months: 4 data collections during the study (baseline, 12 months, 18 months, 24 months)
  The change in incidence of Patient Falls during the study will be investigated by use of repeated measures. The patterns of change between baseline, 12 months, 18 months, and 24 months will be evaluated.
  The data will be collected from the patient's medical file. The timeframe for registration is admission on the ward until discharge from the ward. Any patient falls during the patient's stay on the ward will registered.
Change in Unnecessary New Intravenous Drips | 24 months: 4 data collections during the study (baseline, 12 months, 18 months, 24 months)
  The change in incidence of Unnecessary New Intravenous Drips during the study will be investigated by use of repeated measures. The patterns of change between baseline, 12 months, 18 months, and 24 months will be evaluated.
  The data will be collected from the patient's medical file. The timeframe for registration is from admission on the ward until discharge from the ward with a maximum of 30 days. Newly placed intravenous drips without explicit physician indication will be registered.
Change in Length of Stay | 24 months: 4 data collections during the study (baseline, 12 months, 18 months, 24 months)
  The change in Length of Stay during the study will be investigated by use of repeated measures. The patterns of change between baseline, 12 months, 18 months, and 24 months will be evaluated.
  The data will be collected from the patient's medical file. The total length of stay on the ward will be registered.
Change in Unplanned Readmission | 24 months: 4 data collections during the study (baseline, 12 months, 18 months, 24 months)
  The change in incidence of Unplanned Readmissions during the study will be investigated by use of repeated measures. The patterns of change between baseline, 12 months, 18 months, and 24 months will be evaluated.
  The data will be collected from the patient's medical file. Readmissions within 30 days in the same hospital will be registered.
Change in Pain | 24 months: 4 data collections during the study (baseline, 12 months, 18 months, 24 months)
  The change in Pain scores during the study will be investigated by use of repeated measures. The patterns of change between baseline, 12 months, 18 months, 24 months will be evaluated.
  The data will be collected from the patient's medical file. The timeframe for registration is from admission on the ward until discharge from the ward. The first pain score after the nurse shift report will be registered each day.
Change in Duration of the shift report | 24 months: 4 data collections during the study (baseline, 12 months, 18 months, 24 months)
  The change in the Duration of the Shift Report during the study will be investigated by use of repeated measures. The patterns of change between baseline, 12 months,18 months, and 24 months will be evaluated.
  Thirteen shift reports will be recorded during each data collection point. Based on the recordings, the duration of the shift report will be calculated.
Feasibility | 12 months: 1 data collection (12 months)
  The data concerning the experienced Feasibility of BSR will be collected by use of individual, semi-structured interviews (patients) and semi-structured focus group interviews (nurses) using an interview guide. The data will be collected at 12 months.
Applicability | 12 months: 1 data collection (12 months)
  The data concerning the experienced Applicability of BSR will be collected by use of individual, semi-structured interviews (patients) and semi-structured focus group interviews (nurses) using an interview guide. The data will be collected at 12 months.
Meaningfulness | 12 months: 1 data collection (12 months)
  The data concerning the experienced Meaningfulness of BSR will be collected by use of individual, semi-structured interviews (patients) and semi-structured focus group interviews (nurses) using an interview guide. The data will be collected at 12 months.
Change in Intervention Fidelity | 24 months: 2 data collections during the study(between 12 months and 18 months; between 18 months and 24 months)
  The change in Intervention Fidelity during the study will be investigated by use of repeated measures. The patterns of change will be evaluated.
  The data will be collected by use of non-participating observations. A checklist will be used. During each period (12 months until 18 months / 18 months until 24 months) 20 non-participating observations on each ward will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Van Hecke, MSc, PhD, Principal Investigator — Ghent University/Ghent University Hospital; Kristof Eeckloo, LMM, PhD, Principal Investigator — Ghent University/Ghent University Hospital; Wim Van Biesen, MD, PhD, Principal Investigator — Ghent University/Ghent University Hospital
Locations (8):
- Belgium (8):
  - AZ Sint-Jan, Bruges
  - AZ Alma, Eeklo
  - AZ Sint-Lucas, Ghent
  - Ghent University Hospital, Ghent
  - AZ Virge Jessa, Hasselt
  - AZ Groeninge, Kortrijk
  - AZ Lokeren, Lokeren
  - AZ Oudenaarde, Oudenaarde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson CD, Mangino RR. Nurse shift report: who says you can't talk in front of the patient? Nurs Adm Q. 2006 Apr-Jun;30(2):112-22. doi: 10.1097/00006216-200604000-00008. PMID 16648723
- [Background] Cairns LL, Dudjak LA, Hoffmann RL, Lorenz HL. Utilizing bedside shift report to improve the effectiveness of shift handoff. J Nurs Adm. 2013 Mar;43(3):160-5. doi: 10.1097/NNA.0b013e318283dc02. PMID 23425914
- [Background] Evans D, Grunawalt J, McClish D, Wood W, Friese CR. Bedside shift-to-shift nursing report: implementation and outcomes. Medsurg Nurs. 2012 Sep-Oct;21(5):281-4, 292. PMID 23243785
- [Background] Gonzalo JD, Wolpaw DR, Lehman E, Chuang CH. Patient-centered interprofessional collaborative care: factors associated with bedside interprofessional rounds. J Gen Intern Med. 2014 Jul;29(7):1040-7. doi: 10.1007/s11606-014-2817-x. Epub 2014 Mar 11. PMID 24615186
- [Background] Gregory S, Tan D, Tilrico M, Edwardson N, Gamm L. Bedside shift reports: what does the evidence say? J Nurs Adm. 2014 Oct;44(10):541-5. doi: 10.1097/NNA.0000000000000115. PMID 25208269
- [Background] Griffin SJ, Kinmonth AL, Veltman MW, Gillard S, Grant J, Stewart M. Effect on health-related outcomes of interventions to alter the interaction between patients and practitioners: a systematic review of trials. Ann Fam Med. 2004 Nov-Dec;2(6):595-608. doi: 10.1370/afm.142. PMID 15576546
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America. Crossing the Quality Chasm: A New Health System for the 21st Century. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222274/ PMID 25057539
- [Background] Longtin Y, Sax H, Leape LL, Sheridan SE, Donaldson L, Pittet D. Patient participation: current knowledge and applicability to patient safety. Mayo Clin Proc. 2010 Jan;85(1):53-62. doi: 10.4065/mcp.2009.0248. PMID 20042562
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M. Developing and evaluating complex interventions: the new Medical Research Council guidance. Int J Nurs Stud. 2013 May;50(5):587-92. doi: 10.1016/j.ijnurstu.2012.09.010. Epub 2012 Nov 15. No abstract available. PMID 23159157
- [Background] Smeulers M, Lucas C, Vermeulen H. Effectiveness of different nursing handover styles for ensuring continuity of information in hospitalised patients. Cochrane Database Syst Rev. 2014 Jun 24;2014(6):CD009979. doi: 10.1002/14651858.CD009979.pub2. PMID 24957503
- [Background] Wakefield DS, Ragan R, Brandt J, Tregnago M. Making the transition to nursing bedside shift reports. Jt Comm J Qual Patient Saf. 2012 Jun;38(6):243-53. doi: 10.1016/s1553-7250(12)38031-8. PMID 22737775
- [Derived] Malfait S, Eeckloo K, Van Opdorp L, Van Biesen W, Van Hecke A. The impact of bedside handovers on relevant clinical indicators: A matched-controlled multicentre longitudinal study. J Adv Nurs. 2020 Aug;76(8):2104-2112. doi: 10.1111/jan.14406. Epub 2020 May 25. PMID 32347554